CLINICAL TRIAL: NCT03816943
Title: The Influence of Communication After Placement of Orthodontic Fixed Appliances on Pain, Anxiety and Oral Health Quality of Life Among Malaysian Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Yasmin Kamarudin, Principle investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RF004E-2018
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Orthodontic Pain
Keywords: fixed appliances; orthodontics; quality of life; anxiety; pain; instant messaging; telephone call
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — CD56 Antigen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): control group with no intervention
- Whatsapp (Experimental): intervention group receiving a Whatsapp instant text message with encouraging words after bond up of fixed appliances
  Interventions: Behavioral: Whatsapp
- Call (Experimental): intervention group receiving a phone cal with encouraging words after bond up of fixed appliances
  Interventions: Behavioral: Call

INTERVENTIONS:
Behavioral: Whatsapp — a WhatsApp message with encouraging words will be sent after bond up
  Arms: Whatsapp
Behavioral: Call — a telephone call will be made after bond up to provide encoring words
  Arms: Call

SUMMARY:
Assessing the influence of a telephone call or Whatsapp instant text message post bond up of fixed appliances on Pain Visual Analogue Scores, State-Trait Anxiety and Oral Health Quality of Life

DETAILED DESCRIPTION:
Methodology

Sample 250 new orthodontic patients that meet the research criteria, will be randomly divided into 3 groups (Group 1: Phone call, Group 2: WhatsApp message, Group 3: Control).

Intervention During the bond up appointment, all participants will receive the same advice on pain management. The control group (Group 3) will receive no post bond up intervention whereas the remaining two groups will either receive a single instant text message via WhatsApp (Group 2) or a telephone call (Group 1) 4-7 hours after bond up to provide pain advice, motivation and reassurance. No further message or phone call will be carried out unless the phone call group is unable to be contacted within the 4-7 hour time frame. In this instance, a second phone call will be attempted within 24 hours. The timing of the intervention is based on studies which suggest that pain starts approximately after 4 hours and peaks at 24 hours.

Questionnaires

During the duration of the study, all patients will be required to complete three separate online questionnaires at various time points over a 7-day period. The questionnaires include:

1. Self-reported pain which consists of a Visual Analog Scale (VAS) and a question on analgesic consumption
2. Anxiety questionnaire using the state scale of the Spielberger State-Trait Anxiety Inventory (STAI)
3. Oral health related quality of life using the Oral Health Impact Profile-14

The questionnaires will need to be completed prior to bond up to serve as base line records (T0) and again 4 hours post bonding (T1) followed by daily for the next 7 days at the same time (T2, T3....T7). All questionnaires will be completed online to facilitate easier submission. A link to the online survey will be emailed directly to the patients daily as each patient will have to complete the survey at different times depending on the timing of their bond up appointment.

An additional pain questionnaire (TE) will be completed prior to extractions to make sure pain levels have returned to normal during the bond up appointment.

Statistical analysis Statistical Package for Social Sciences (SPSS) will be used to analyse the data.

To reduce risk of bias, the clinician, patient and the statistician will be blinded to the intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* New patients requiring fixed preadjusted appliances in both arches
* Age ≥ 16 years old
* Patients of Mongoloid ethnicity
* Patients with access to a cellular phone with Whatsapp instant messaging app
* Patients with access to internet services and email account for questionnaire completion
* Patients with partial bond up e.g delayed bond up of lower incisors or upper laterals

Exclusion Criteria:

* History of reported chronic use of analgesic medication
* History of chronic pain related pathology or disease
* History of previous fixed orthodontic intervention
* Patients that have recently had teeth extracted less than 2 weeks prior to bond up
* Patients requiring bond of both arches on separate days
* Syndromic patients

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
change in pain (VAS) | every day for 1 week post bond up
  measure daily change in pain post bonding of fixed appliances using a 10mm pain visual analogue scale. 0mm = no pain and 100mm = worst pain imaginable

SECONDARY OUTCOMES:
Change in Anxiety (STAI) | everyday for 1 week post bond up. It consists of 40 statements which require the participant to rate using a 4 point likert scale.Total scores can range between 40 to 160. Higher scores indicate increased anxiety .
  Measure daily change in anxiety post bonding of fixed appliances using the State-Trait Anxiety Inventory (STAI)

OTHER OUTCOMES:
Change in Quality of life (OHIP-16) | everyday for 1 week post bond up
  Measure daily change in Oral health quality of life using the modified short Malay version of the Oral Health Impact Profile (OHIP-16M).It consists of a Likert scale and coded as: 1=never, 2=hardly ever, 3=occasionally, 4=fairly often, and 5=very often. The OHIP-16[M] scores range from 16 to 80, where 16 indicates no impact and 80 indicates the worst impact of one's oral health on QOL.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartlett BW, Firestone AR, Vig KW, Beck FM, Marucha PT. The influence of a structured telephone call on orthodontic pain and anxiety. Am J Orthod Dentofacial Orthop. 2005 Oct;128(4):435-41. doi: 10.1016/j.ajodo.2004.06.033. PMID 16214624
- [Background] Cozzani M, Ragazzini G, Delucchi A, Barreca C, Rinchuse DJ, Servetto R, Calevo MG, Piras V. Self-reported pain after orthodontic treatments: a randomized controlled study on the effects of two follow-up procedures. Eur J Orthod. 2016 Jun;38(3):266-71. doi: 10.1093/ejo/cjv032. Epub 2015 Jun 11. PMID 26070922
- [Background] Keith DJ, Rinchuse DJ, Kennedy M, Zullo T. Effect of text message follow-up on patient's self-reported level of pain and anxiety. Angle Orthod. 2013 Jul;83(4):605-10. doi: 10.2319/091812-742.1. Epub 2012 Dec 4. PMID 23210546
- [Background] Mansor N, Saub R, Othman SA. Changes in the oral health-related quality of life 24 h following insertion of fixed orthodontic appliances. J Orthod Sci. 2012 Oct;1(4):98-102. doi: 10.4103/2278-0203.105880. PMID 24987635
- [Background] Ngan P, Kess B, Wilson S. Perception of discomfort by patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1989 Jul;96(1):47-53. doi: 10.1016/0889-5406(89)90228-x. PMID 2750720